CLINICAL TRIAL: NCT07180849
Title: Comparing the Antiplaque Efficacy of Titania Nanoparticle Infused Fluoride Varnish vs Conventional Fluoride Varnish in Fixed Orthodontic Patients-A Triple Blind Randomised Controlled Trial.
Brief Title: Comparing the Antiplaque Effects of Novel Titania Nanoparticle Infused Fluoride Varnish vs Conventional Fluoride Varnish in Fixed Orthodontic Patients.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Pakistan Institute of Medical Sciences (Other Government)
Responsible Party: Principal Investigator, Afifa Fahim, Principal Investigator, Pakistan Institute of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: SOD/ERB/2025/91
Record Dates: First submitted 2025-09-12; First posted 2025-09-18 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Dental Plaque Accumulation; Nanoparticles; Fluoride Varnishes

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): Group A will receive topical application of conventional fluoride varnish.
  Interventions: Procedure: Fluoride varnish
- Group B (Experimental): Group B will receive topical application of titania nanoparticle infused varnish.
  Interventions: Procedure: Novel titania nanoparticle infused fluoride varnish

INTERVENTIONS:
Procedure: Fluoride varnish — Group A will receive conventional fluoride varnish for antiplaque effects.Plaque will be assessed quantitatively by modified plaque index.
  Arms: Group A
Procedure: Novel titania nanoparticle infused fluoride varnish — Group B will receive topical application of titania nanoparticle infused fluoride varnish for antiplaque effects.Plaque will be assessed quantitatively by modified plaque index.
  Arms: Group B

SUMMARY:
In this study the investigators aimed to explore the antibiofilm effect of fluoride varnish loaded with titania nanoparticles synthesized from moringa oleifera leaves extract vs conventional fluoride varnish in multibracket fixed orthodontic patients.

ELIGIBILITY:
Inclusion criteria:

* Patients planned for fixed orthodontic treatment.
* Patients within age group 16-30 years.
* Patient with no history of previous orthodontic treatment.
* Patients with no active periodontal diseases.

Exclusion criteria:

* Patient undergoing any antibiotic therapy.
* Patients with any craniofacial abnormality.
* Patient with mixed dentition

Ages: 16 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-11 (Estimated); Primary Completion 2027-07 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
To compare the plaque inhibitory effect of titania nanoparticle infused fluoride varnish and conventional fluoride varnish in fixed orthodontic patients. | 6 months
  Plaque will be assessed quantitatively by modified plaque index.

SECONDARY OUTCOMES:
To measure plaque bacterial load and pH following application of titania nanoparticle infused and conventional fluoride varnish in fixed orthodontic patients. | 6 months
  Bacterial colonies will be morphologically identified and counted as Colony Forming Units (CFU) using a colony counting grid.

CONTACTS AND LOCATIONS:
Locations (1):
- Pakistan Institute of Medical Sciences, Islamabad, Pakistan